CLINICAL TRIAL: NCT01425255
Title: Prospective Exploratory Study Evaluating Sleep Quality and Sleep-Wake Patterns in Parents of Children With Type 1 Diabetes Before and Several Weeks After Initiating Using RT-CGM of Their Children.
Brief Title: The Impact of Continuous Glucose Monitoring Use on Sleep in Parents of Children With Type 1 Diabetes Mellitus
Status: Withdrawn | Type: Observational
Why Stopped: Enrollment finished and a paper was published.
Sponsor: Wolfson Medical Center (Other Government)
Collaborators: Tel Aviv Medical Center (Other); Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, zohar landau, Head of Pediatric Endocrinology Service, Wolfson Medical Center
Other Study IDs: 0077-11-WOMC
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2011-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Sleep quality; Parents
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parents of children with Type 1 diabetes: before and several weeks after initiating using RT-CGM of their children.

SUMMARY:
The purpose of this prospective exploratory study is to compare sleep quality and sleep-wake patterns in parents of children with type 1 diabetes (T1D) before and several weeks after initiating using real-time continuous glucose monitoring (RT-CGM) of their children.

DETAILED DESCRIPTION:
Few weeks before scheduled initiation of RT-CGM use of a child with T1D, the 'dominant parent' (the main caregiver during the nighttime in the family) will obtain an informed consent. This will be done during a routine visit in the diabetes clinic. The participants will complete a sleep quality questionnaire (PSQI) and instructions on care of the actigraph and how to keep complete the daily sleep diary will be given. The participants will be instructed to wear the actigraph for 7 consequences nights. Four to eight weeks after initiation of RT-CGM use, the 'dominant parent' will be asked to wear the actigraph for 7 consequences nights and to complete the sleep quality questionnaire and the daily sleep diary.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children up to 16 years old with type 1 diabetes

Exclusion Criteria:

* Either the child or parent had obstructive sleep apnea, narcolepsy, or restless legs syndrome.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Juvenile Diabetes Clinics
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
sleep quality | 1 year
  Actigraphy:
  Sleep Diary:During the weeks participants will wear the actigraph, they will be asked to rate their previous nights' sleep using a very short questionnaire.
  Pittsburgh Sleep Quality Index (PSQI):

SECONDARY OUTCOMES:
Glycemic control | one year
  1. HbA1c level
  2. Mean blood glucose level:
  3. Number of severe hypoglycemic episodes and diabetic ketoacidoacidosis episodes

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Landau, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- E. Wolfson Medical Center, Holon, Israel